CLINICAL TRIAL: NCT02626572
Title: Efficacy and Safety of 3 Doses of S47445 Versus Placebo in Patients With Alzheimer's Disease at Mild to Moderate Stages With Depressive Symptoms. A 24-week International, Multi-centre, Randomized, Double-blind, Placebo-controlled Phase II Study in Monotherapy Followed by an Optional 28-week Extension Period in Co-administration With Donepezil.
Brief Title: Efficacy and Safety of 3 Doses of S47445 Versus Placebo in Patients With Alzheimer's Disease at Mild to Moderate Stages With Depressive Symptoms
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut de Recherches Internationales Servier (Other)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CL2-47445-011; 2014-001519-38 (EudraCT Number)
Record Dates: First submitted 2015-11-04; First posted 2015-12-10 (Estimated); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- S47445 5mg (Experimental)
  Interventions: Drug: S47445 5mg
- S47445 15mg (Experimental)
  Interventions: Drug: S47445 15mg
- S47445 50mg (Experimental)
  Interventions: Drug: S47445 50mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: S47445 5mg — S47445 5 mg tablets taken orally once a day during breakfast, starting the day after inclusion visit and ending the day of the W024 visit (main period) or starting the day after inclusion visit and ending the day of the W052 visit (period including main period and optional extension period).
  Arms: S47445 5mg
Drug: S47445 15mg — S47445 15 mg tablets taken orally once a day during breakfast, starting the day after inclusion visit and ending the day of the W024 visit (main period) or starting the day after inclusion visit and ending the day of the W052 visit (period including main period and optional extension period).
  Arms: S47445 15mg
Drug: S47445 50mg — S47445 50 mg tablets taken orally once a day during breakfast, starting the day after inclusion visit and ending the day of the W024 visit (main period) or starting the day after inclusion visit and ending the day of the W052 visit (period including main period and optional extension period).
  Arms: S47445 50mg
Drug: Placebo — Placebo tablets taken orally once a day during breakfast, starting the day after inclusion visit and ending the day of the W024 visit (main period) or starting the day after inclusion visit and ending the day of the W052 visit (period including main period and optional extension period).
  Arms: Placebo

SUMMARY:
The purpose of this trial is to assess the efficacy and safety of S47445 versus placebo in patients with Alzheimer's disease at mild to moderate stages with depressive symptoms. An optional 28-week extension period will be performed to evaluate safety/tolerance and efficacy of S47445 in co-administration with donepezil.

ELIGIBILITY:
Inclusion Criteria:

* Out-patients
* Able to perform neuropsychological tests
* Have a responsible informant
* DSM-IV-TR criteria for Dementia of the Alzheimer's Disease Type
* Mini mental State Examination (MMSE) = 15-24 both inclusive
* National Institute of Mental Health (NIMH) provisional criteria for depression in AD (NIMH-dAD)
* Cornell Scale for Depression in Dementia total score > or = 8
* Patients who have never been treated with AD treatments or patients who have stopped AD treatment whatever the reason
* Patients either not currently treated with an antidepressant or patients being treated with an antidepressant at the recommended dose for at least 8 weeks without clinical efficacy, who can stop this treatment according to the investigator's opinion.

Exclusion Criteria:

* Patients not able to read or write
* Patients having participated in a study testing disease modifying therapy for AD, or in another study with administration of investigational drug or device within the previous 3 months prior to selection visit
* Depressive symptoms that, in investigator's judgment, are clearly due to a medical condition other than AD, or are a direct result of non-mood related dementia symptoms
* History of epilepsy or solitary seizure
* Medical history of Major Depressive Disorder more than 3 years before onset of the disease, treated with antidepressive drugs or electroconvulsive therapy
* Severe or unstable disease of any type that could interfere with safety and efficacy assessments
* Alcohol abuse or drug abuse or addiction, as judged by the clinician (excluding nicotine)
* Clinically relevant lactose intolerance
* Antidepressant treatment not stopped for at least 3 weeks before inclusion
* Significant worsening of depressive symptoms or high suicidal risk according to investigator's judgment
* For optional extension phase: medically instable Chronic Obstructive Pulmonary Disease and asthma, known hypersensitivity to donepezil hydrochloride or piperidine derivatives

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2015-02; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline on 11-item ADAS-Cog | 24 weeks of treatment
  Cognition criterion

SECONDARY OUTCOMES:
Activities of Daily Living: Disability Assessment for Dementia (DAD) | baseline, week 12, week 24 and week 52
  Key secondary efficacy criterion
Cognition: 13-item ADAS-Cog | baseline, week 4, week 12, week 24, week 38 and week 52
  Other secondary efficacy criteria
Cognition: Mini-Mental State Examination (MMSE) | baseline, week 12, week 24 and week 52
  Other secondary efficacy criteria
Depressive symptoms: Cornell Scale for Depression in Dementia (CSDD) | baseline, week 4, week 12, week 24, week 38 and week 52
  Other secondary efficacy criteria
Behavioural signs and symptoms: Neuropsychiatric Inventory (NPI) | baseline, week 4, week 12, week 24 and week 52
  Other secondary efficacy criteria
Global Clinic Assessment of Change: Alzheimer's Disease Cooperative Studies-Clinical Global Impression of Change (ADCS-CGIC) | baseline, week 24 and week 52
  Other secondary efficacy criteria
Functionality: Gait task (GT), measure of speed of walking (unit= meters/ seconds) | baseline, week 4, week 12, week 24, week 38 and week 52
  Other secondary efficacy criteria
Adverse events | through study completion, an average of 1 year
  Safety criterion
Vital signs: heart rate | baseline, week 4, week 12, week 24, week 38 and week 52
  Safety criterion
Vital signs: body temperature | baseline, week 4, week 12, week 24, week 38 and week 52
  Safety criterion
Vital signs: blood pressure | baseline, week 4, week 12, week 24, week 38 and week 52
  Safety criterion
Vital signs: body weight | baseline, week 12, week 24, week 38 and week 52
  Safety criterion
12-lead ECG | baseline, week 4, week 12, week 24, week 38 and week 52
  Safety criterion
Biological laboratory parameters: number of participants with abnomal laboratory values | baseline, week 4, week 12, week 24, week 38 and week 52
  Safety criterion
Cornell Scale for Depression in Dementia (CSDD, suicide item - item 16) | baseline, week 4, week 12, week 24, week 28, week 38 and week 52
  Safety criterion

CONTACTS AND LOCATIONS:
Locations (78):
- Brazil (7):
  - Trial Tech Tecnologia em Pesquisa com Medicamentos, Curitiba
  - Hospital Universitario Walter Cantidio, Fortaleza
  - Clinilive - Centro de Pesquisas Clinicas, Maringá
  - Hospital das Clinicas de Porto Alegre, Porto Alegre
  - Hospital Oswaldo Cruz, Recife
  - Instituto Américo Bairral de Psiquiatria, Centro de Pesquisa, São Paulo
  - UNIFESP - Universidade Federal de Sao Paulo, São Paulo
- Bulgaria (5):
  - UMHAT Sveti Georgi, Plovdiv
  - Medical University of Sofia, Aleksandrovska hospital, Sofia
  - National Hospital of Cardiology, Sofia
  - University Hospital Sveti Naum, Clinic of Neurology, Sofia
  - MHAT Sveta Marina, Varna
- Chile (5):
  - Clínica Oriente, Antofagasta
  - Biomedica Research Group, Santiago
  - Especialidades Medicas LYS, Santiago
  - Hospital Santiago Oriente, Santiago
  - Private practice, Santiago
- Czechia (6):
  - Saint Anne s.r.o. Psychiatricka ambulance, Brno
  - Brain-Soultherapy s.r.o., Kladno
  - Bialbi s.r.o., Litoměřice
  - AD71 s.r.o. Psychiatricka ambulance - Sudkova, Prague
  - CLINTRIAL s.r.o., Prague
  - FORBELI s.r.o., Neurologicka ambulance, Prague
- Germany (8):
  - Klinikum Altenburger Land GmbH Neurologische Klinik, Altenburg
  - Neuropsychiatrisches Facharztzentrum Stiepel, Bochum
  - Universitaetsklinikum des Saarlandes, Klinik für Psychiatrie und Psychotherapie, Homburg / Saar
  - ISPG Institut für Studien zur Psychischen Gesundheit, Mannheim
  - Pharmakologisches Studienzentrum Chemnitz GmbH, Mittweida
  - Somni Bene, Institut fuer Medizinische Forschung und Schlafmedizin Schwerin GmbH, Schwerin
  - Universitaetsklinik ULM, Poliklinik Neurologie, Ulm
  - Private practice, Westerstede
- Hungary (10):
  - Semmelweis Egyetem Neurologiai Klinika, Budapest
  - Kenezy Gyula Korhaz es Rendelointezet, Debrecen
  - Vaszary Kolos Korhaz Esztergom Neurologiai Osztaly, Esztergom
  - Petz Aladar Megyei Oktato Korhaz Pszihiatriai, Mentalhygienes es Addiktologiai Osztaly, Győr
  - Private practice, Kalocsa
  - B-A-Z Megyei Korhaz es Egyetemi Oktato Korhaz Stroke, Er- es Neurologiai, Toxikologiai Osztaly, Miskolc
  - Josa Andras Oktatokorhaz Pszihiatriai Osztaly, Nyíregyháza
  - Pecsi Tudomanyegyetem, Klinikai Kozpont Pszich. es Pszichoter. Klinika, Pécs
  - Szent-Gyorgyi Albert Klinikai Kozpont Pszichiatriai Klinika, Szeged
  - Fejer Megyei Szent Gyorgy Egyetemi Oktato Korhaz Pszichiatriai Osztaly, Székesfehérvár
- Japan (9):
  - Memory Clinic Ochanomizu, Bunkyō City
  - Showakai Clinic, Kagoshima
  - Rainbow & Sea Hospital, Karatsu-shi
  - Kokan Clinic, Kawasaki-shi
  - Social Medical Corporation Kojunkai Daido Hospital, Nagoya
  - Nakano General Hospital, Nakano
  - Private practice, Saitama-shi
  - Private practice, Setagaya-ku
  - Seishinkai Okehazama Hospital, Toyoake-shi
- Mexico (4):
  - Instituto Biomedico de Investigacion, Aguascalientes
  - Centro de Estudios Clinicos Y Especialidades Medicas Sc, Monterrey
  - Hospital Universitario de Nuevo León, Nuevo León
  - University Hospital of Saltillo, Saltillo
- Poland (6):
  - Nzoz Centrum Kultury, Higieny I Zdrowia Psychicznego, Bydgoszcz
  - Krakowska Akademia Neurologii Centrum Neurologii Klinicznej, Krakow
  - NZOZ Neuromed M. i M. Nastaj Sp. Partnerska, Lublin
  - SENIOR Poradnia Psychogeriatryczna, Sopot
  - Osrodek Alzheimerowski Sp. z o.o., Ścinawa
  - Centrum Medyczne Neuroprotect, Warsaw
- Russia (8):
  - Interregional Clinico-Diagnostical Centre, Kazan'
  - First Moscow State Medical University n.a.I.M. Sechenov Clinic of Neurology, Moscow
  - Scientific Center of Mental Health Sect of AD and associated disord. Dpt of gerontopsychiatry, Moscow
  - Scientific Center of Mental Health Sect of psychosis of elderly ages Dpt of gerontopsychiatry, Moscow
  - City geriatric medico-social centre, Saint Petersburg
  - Medical Military Academy n.a.S.M.Kirov, Saint Petersburg
  - Psychoneuropathology Dispensary N 10, Saint Petersburg
  - Co Ltd "LION-MED", Voronezh
- Slovakia (3):
  - Private practice, Bratislava
  - INVESTA, spol. s r. o. Psychiatricka ambulancia, Košice
  - NsP Svatej Barbory Psychiatricke oddelenie, Rožňava
- South Africa (7):
  - Iatros International, Bloemfontein
  - Flexivest Fourteen Research Centre, Cape Town
  - Umhlanga Hospital, Durban
  - Excellentis Clinical Trial Consultants, George
  - Apollo Clinical Research, Johannesburg
  - Denmar Hospital, Pretoria
  - Somerset West Trial Centre, Somerset West

IPD SHARING:
Plan to Share IPD: Yes
Researchers can ask for a study protocol, patient-level and/or study-level clinical trial data including clinical study reports (CSRs).
  They can ask all interventional clinical studies:
  * submitted for new medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * Where Servier or an affiliate are the Marketing Authorization Holders (MAH). The date of the first Marketing Authorization of the new medicine (or the new indication) in one of the EEA Member States will be considered within this scope.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorisation in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: http://clinicaltrials.servier.com

REFERENCES:
- [Result] Bernard K, Gouttefangeas S, Bretin S, Galtier S, Robert P, Holthoff-Detto V, Cummings J, Pueyo M. A 24-week double-blind placebo-controlled study of the efficacy and safety of the AMPA modulator S47445 in patients with mild to moderate Alzheimer's disease and depressive symptoms. Alzheimers Dement (N Y). 2019 Jun 24;5:231-240. doi: 10.1016/j.trci.2019.04.002. eCollection 2019. PMID 31297437